CLINICAL TRIAL: NCT02115100
Title: Treatment of Atrial Fibrillation in Patients With High Sympathetic Activity by Pulmonary Vein Isolation in Combination With Renal Denervation or Pulmonary Vein Isolation Only; an International Randomized, Controlled Trial
Brief Title: Treatment of Atrial Fibrillation in Patients by Pulmonary Vein Isolation in Combination With Renal Denervation or Pulmonary Vein Isolation Only
Acronym: ASAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diagram B.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9206
Record Dates: First submitted 2014-04-10; First posted 2014-04-15 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Out of Range Hypertension; Signs of Sympathetic Overdrive
Keywords: Paroxysmal atrial fibrillation; Persistent atrial fibrillation; Out of range hypertension; Signs of sympathetic overdrive
MeSH Terms: conditions — Atrial Fibrillation | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pulmonary vein+renal artery denervation (Active Comparator): Procedure: pulmonary vein and renal artery denervation
  Interventions: Procedure: procedure
- Pulmonary vein isolation (Active Comparator): Procedure: Pulmonary vein isolation
  Interventions: Procedure: procedure

INTERVENTIONS:
Procedure: procedure — Renal ablation+pulmonary vein isolation OR pulmonary vein isolation only
  Other Names: Renal ablation+pulmonary vein isolation OR pulmonary vein isolation only

SUMMARY:
Prospective, randomized, controlled, multicenter, international clinical trial. The study population consist of patients with paroxysmal or persistent atrial fibrillation with out range hypertension or signs of sympathetic overdrive. Patient will be randomized into one of the following two groups.

group 1 : patients will undergo pulmonary vein isolation, group 2: Patients will undergo pulmonary vein isolation and renal artery denervation.

DETAILED DESCRIPTION:
The target group of patients are subjects ages <65 years, with paroxysmal or persistent atrial fibrillation, who have out of range hypertension (systolic >140 mmHg or >130/80 mmHg in diabetics and patients with chronic renal disease) or signs of sympathetic overdrive. Patients should use at least 2 anti-hypertensive's or should be intolerant for antihypertensive medication.

Atrial fibrillation terminology: If atrial fibrillation recurs more than once but terminates spontaneously within seven days, the term paroxysmal AF is used. This is also used when the episode is less than 48 hours in duration and is terminated with electrical or pharmacological cardioversion. Persistent AF is defined as recurrent AF that is sustained for more than seven days. A patient that is electrically or pharmacologically cardioverted after more than two days is also diagnosed with persistent AF.

After the exclusion of apparent secondary causes of hypertension, patients will be randomized to one of the following interventional treatments:

First arm: PVI (69 patients) Second arm: PVI + RDN (69 patients)

The patient will be treated under conscious sedation or general anesthesia. The control group will consist of patients who undergo PVI alone. The study will be a randomized, controlled trial. The follow up period will be up to one year after the interventional therapy. Patients will be treated clinically and will have regular follow-up at the outpatient clinic of the hospital at which they were treated. If patients receive continuous loop recorders for cardiac rhythm monitoring, this data will be used for the study. The other patients will undergo Holter ECG monitoring at regular intervals during follow-up (at 3, 6 and 12 months after the interventional treatment). During follow-up, the first 3 months after the interventional treatment will be a blanking period, as is common in the ablative therapy of AF (ablations points need to heal, and paroxysms of AF in this period are not associated with therapy failure).

ELIGIBILITY:
Inclusion Criteria:

1. The patient is willing and able to comply with the protocol and has provided written informed consent.
2. The patient falls within the target group resistant hypertension or sympathetic overdrive
3. Patient is an acceptable candidate for renal denervation treatment
4. Patient is < 65 year of age

Exclusion Criteria:

1. Documented left atrial diameter on trans thoracic echocardiography (PLAX > 4.5 cm).
2. Contraindication to chronic anticoagulation therapy or heparin.
3. Previous left heart ablation procedure for AF (atrial fibrillation).
4. Acute coronary syndrome, cardiac surgery, PCI (percutaneous coronary intervention)or stroke within 3 months prior to enrollment.
5. Untreated hypothyroidism or hyperthyroidism.
6. More than grade 1/3 valvular regurgitation and/or significant valve stenosis (modest or severe).
7. LVEF (Left ventricular function) <45% and/or grade 3/4 diastolic dysfunction.
8. Enrollment in another investigational drug or device study.
9. Woman currently pregnant or breastfeeding or not using reliable contraceptive measures during fertile age.
10. Mental or physical inability to participate in the study.
11. Planned cardiovascular intervention.
12. Life expectancy ≤ 12 months.
13. Renal artery stenosis >50% of the arterial lumen, or renal artery lumen

    ≤3 mm.
14. Dual or triple ipsilateral renal artery ostia.
15. Obvious secondary cause of hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2014-03-18 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

PRIMARY OUTCOMES:
Time to first detection of atrial fibrillation > 30 seconds, with the monitoring period starting 3 months after the intervention. | 3 months

SECONDARY OUTCOMES:
A-fib burden during follow-up, expressed in % of the monitoring period, in patients with continuous rhythm monitoring. | 12 months
  The monitoring starts after 3 months
Blood pressure after intervention, and change in blood pressure compared to measurement before the intervention | 3/6/12 months
Blood pressure and heart rate response changes induced by exercise testing | 12 months
Changes in cardiac sympathetic innervation post-intervention compared to measurement before intervention by MIBG in a subset of patients | 12 months
Changes in heart rate variability measures tested by Holter monitoring compared to measurements before the intervention | 12 months
Changes in biomarkers post intervention representing sympathetic tone compared to before the intervention | 12 months
Changes in arterial stiffness measures post intervention ambulatory arterial stiffness index by ambulatory blood pressure monitoring, pulse wave velocity and augmentation index compared to measurement before the intervention | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arif Elvan, MD, PhD, Principal Investigator — Maatschap Cardiologie Isala
Locations (8):
- Netherlands (3):
  - Isala hospital, Zwolle, Overijssel
  - MUMC, Maastricht
  - Radboudumc, Nijmegen
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Fundación Jimenez Díaz, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga

REFERENCES:
- [Derived] Younis A, Steinberg JS. Renal Denervation for Patients With Atrial Fibrillation. Curr Cardiol Rep. 2021 Jul 16;23(9):126. doi: 10.1007/s11886-021-01558-4. PMID 34269911